CLINICAL TRIAL: NCT03540732
Title: Feeding With Indirect Calorimetry and Cycling in the Elderly Intensive Care Patient
Brief Title: Feeding With Indirect Calorimetry and Cycling in the Elderly
Acronym: FICE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017/00573
Record Dates: First submitted 2018-01-31; First posted 2018-05-30 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-06

CONDITIONS: Calorimetry, Indirect; Exercise Therapy; Critical Care; Muscular Atrophy
MeSH Terms: conditions — Muscular Atrophy

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor (in our study, person measuring participants' quadriceps muscle thickness) is blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1. Control (No Intervention): * Standard physiotherapy
  * Empiric formula directed feeding (daily caloric requirement calculated by 25 kcal/kg/day)
- 2. Intervention (Active Comparator): * Up to 60 minutes of cycle ergometry daily in addition to standard physiotherapy sessions.
  * Indirect calorimetry directed feeding (use of indirect calorimetry to calculate daily caloric requirement)
  Interventions: Other: Indirect Calorimetry directed feeding.; Procedure: Cycle Ergometry

INTERVENTIONS:
Other: Indirect Calorimetry directed feeding. — Indirect calorimetry directed feeding (use of indirect calorimetry to calculate daily caloric requirement)
  Arms: 2. Intervention
Procedure: Cycle Ergometry — Up to 60 minutes of cycle ergometry daily in addition to standard physiotherapy sessions.
  Arms: 2. Intervention

SUMMARY:
The aim of this study is to evaluate the effect of early exercise by cycle ergometry and early targeted feeding in reducing muscle atrophy and improve functional outcomes in the older critically ill patient.

DETAILED DESCRIPTION:
Patients admitted to ICU are normally ventilated due to their critical illness and sedated for their comfort. This prolonged immobility from sedation leads to accelerated muscle atrophy and reconditioning when they recover from their critical illness. This leads to further complications from immobility like bed sores, hospital acquired infections, deep vein thrombosis and pulmonary embolisms. Many patients do not return to their pre-illness level of function and require long term care.

Nutrition is frequently hard to assess when patients is in a catabolic state and sedated. There is a loss of appetite if the patient is awake to express it, and if sedated is depended on nasogastric feeding based on caloric empirical formulas invented more than 50 years ago. These formulas also do not accurately take into account exercise physiotherapy which patients will undergo while on ICU. With indirect calorimetry (IC), patients energy requirements can be estimated on a daily basis and can be fed accordingly. The IC is considered the gold standard in many guidelines for nutritional assessments but it is not commonly used due to cost and practical difficulties in measurements. The investigators intend to use the IC based on international recommendations to assess energy requirements daily and feed patients based on the data provided by the IC.

Early rehabilitative type of exercises have been show to increase muscle mass and reduce length of stay in the elderly geriatric population by preventing deconditioning. There is some evidence that this also applies to the ICU population but in a ventilated patient on multiple therapies, this is extremely labour intensive. By utilising the cycle ergometry, this muscle atrophy may be reduced. Interestingly, studies on intensive physiotherapy have not shown to have a dramatic outcome in the elderly ICU population. This could be due to the catabolic rates and the inadequate feeding of a sedated patient who cannot express their hunger or satiety. By using the indirect calorimetry, a more accurate energy expenditure can be estimated and nutrition can be targeted. By combining these 2 therapies, the lengths of stay in hospital can be reduced and functional outcomes improved in this silver population.

The investigators plan to conduct a randomised controlled trial. Participants will be randomised into 2 groups; the intervention and control group. Participants in the control group will receive standard empiric weight based feeding and standard physiotherapy. Participants in the intervention group will undergo daily IC measurements on admission and fed according to the energy expenditure measured by IC. In addition to standard physiotherapy, the participants in the intervention group will undergo cycle ergometry for up to 60 minutes daily. The participants in the intervention group will undergo 14 days of IC and cycle ergometry or until extubation (for IC), whichever is earlier.

During this 14 day period, participants in both groups will undergo twice weekly quadriceps muscle ultrasounds to assess muscle thickness as a surrogate measure of muscle atrophy. After this 14 day period, the investigators will perform regular assessments of functional status (during the ICU/HD stay, on discharge to general ward, and on discharge from hospital). The investigators will also collect demographic and ICU assessment data from medical records.

ELIGIBILITY:
Inclusion Criteria:

1. At least 60 years old
2. Mechanically ventilated within 3 days of ICU admission
3. Expected to be mechanically ventilated for more than 3 days at time of recruitment
4. Able to ambulate with or without a gait aid before hospitalization
5. Able to be enterally fed within 48 hours of ICU admission

Exclusion Criteria:

1. Unable to follow commands at baseline before hospital admission (e.g. Severe dementia)
2. Acute condition where cycling is a contraindication (e.g. leg fracture)
3. Not expected to survive the subsequent 48 hours
4. Body habitus unable to fit the cycle ergometry
5. Patients at high risk of refeeding (i.e. NUTRIC score >= 5): malnourished patients with anorexia nervosa, chronic malabsorption syndromes, chronic alcoholism, or patients with massive weight loss.
6. Extremes of BMI: i.e. BMI < 16 or > 30
7. Liver failure
8. Cycling exemptions precluding cycling within the first 4 days of mechanical ventilation
9. Requirement for inspired oxygen content (FiO2) greater than 0.8
10. Expected to be on renal replacement therapy for longer than 12 hours per session
11. PEEP > 15mmHg
12. Air leaks through chest drains
13. Palliative goals of care or limitation of treatment established by the CARE form
14. Readmissions to ICU

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-11-06 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in quadriceps muscle thickness | Change in thickness of quadriceps muscle (as assessed by ultrasound scanning) over the first 2 weeks of study.
  Change in quadriceps muscle thickness

SECONDARY OUTCOMES:
MRC-ss | On discharge from ICU, up to 1 year from recruitment.
  Measurement of functional outcome.
MRC-ss | 14 days after recruitment
  Measurement of functional outcome.
MRC-ss | On discharge from hospital, up to 1 year from recruitment.
  Measurement of functional outcome.
FSS-ICU | On discharge from ICU, up to 1 year from recruitment.
  Measurement of functional outcome.
FSS-ICU | 14 days after recruitment
  Measurement of functional outcome.
FSS-ICU | On discharge from hospital, up to 1 year from recruitment.
  Measurement of functional outcome.
CPax | On discharge from ICU, up to 1 year from recruitment.
  Measurement of functional outcome.
CPax | 14 days after recruitment
  Measurement of functional outcome.
CPax | On discharge from hospital, up to 1 year from recruitment.
  Measurement of functional outcome.
Quadriceps strength and hand grip strength | On discharge from ICU, up to 1 year from recruitment.
  Measured with dynamometer.
Quadriceps strength and hand grip strength | 14 days after recruitment
  Measured with dynamometer.
Quadriceps strength and hand grip strength | On discharge from hospital, up to 1 year from recruitment.
  Measured with dynamometer.
Length of Stay in ICU | Day of discharge from ICU, up to 1 year from recruitment.
  Length of Stay in ICU
Length of hospital stay | Day of discharge from hospital, up to 1 year from recruitment.
  Length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Will NH Loh, MBBS, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Health System, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Puthucheary ZA, Rawal J, McPhail M, Connolly B, Ratnayake G, Chan P, Hopkinson NS, Phadke R, Dew T, Sidhu PS, Velloso C, Seymour J, Agley CC, Selby A, Limb M, Edwards LM, Smith K, Rowlerson A, Rennie MJ, Moxham J, Harridge SD, Hart N, Montgomery HE. Acute skeletal muscle wasting in critical illness. JAMA. 2013 Oct 16;310(15):1591-600. doi: 10.1001/jama.2013.278481. PMID 24108501
- [Background] Wei X, Day AG, Ouellette-Kuntz H, Heyland DK. The Association Between Nutritional Adequacy and Long-Term Outcomes in Critically Ill Patients Requiring Prolonged Mechanical Ventilation: A Multicenter Cohort Study. Crit Care Med. 2015 Aug;43(8):1569-79. doi: 10.1097/CCM.0000000000001000. PMID 25855901
- [Background] Wichansawakun S, Meddings L, Alberda C, Robbins S, Gramlich L. Energy requirements and the use of predictive equations versus indirect calorimetry in critically ill patients. Appl Physiol Nutr Metab. 2015 Feb;40(2):207-10. doi: 10.1139/apnm-2014-0276. Epub 2014 Oct 27. PMID 25610953
- [Background] Parry SM, Huang M, Needham DM. Evaluating physical functioning in critical care: considerations for clinical practice and research. Crit Care. 2017 Oct 4;21(1):249. doi: 10.1186/s13054-017-1827-6. PMID 28978333
- [Background] Reid CL. Poor agreement between continuous measurements of energy expenditure and routinely used prediction equations in intensive care unit patients. Clin Nutr. 2007 Oct;26(5):649-57. doi: 10.1016/j.clnu.2007.02.003. Epub 2007 Apr 6. PMID 17418917
- [Background] Singer P, Anbar R, Cohen J, Shapiro H, Shalita-Chesner M, Lev S, Grozovski E, Theilla M, Frishman S, Madar Z. The tight calorie control study (TICACOS): a prospective, randomized, controlled pilot study of nutritional support in critically ill patients. Intensive Care Med. 2011 Apr;37(4):601-9. doi: 10.1007/s00134-011-2146-z. Epub 2011 Feb 22. PMID 21340655
- [Background] Kho ME, Molloy AJ, Clarke FJ, Ajami D, McCaughan M, Obrovac K, Murphy C, Camposilvan L, Herridge MS, Koo KK, Rudkowski J, Seely AJ, Zanni JM, Mourtzakis M, Piraino T, Cook DJ; Canadian Critical Care Trials Group. TryCYCLE: A Prospective Study of the Safety and Feasibility of Early In-Bed Cycling in Mechanically Ventilated Patients. PLoS One. 2016 Dec 28;11(12):e0167561. doi: 10.1371/journal.pone.0167561. eCollection 2016. PMID 28030555
- [Background] Seymour JM, Ward K, Sidhu PS, Puthucheary Z, Steier J, Jolley CJ, Rafferty G, Polkey MI, Moxham J. Ultrasound measurement of rectus femoris cross-sectional area and the relationship with quadriceps strength in COPD. Thorax. 2009 May;64(5):418-23. doi: 10.1136/thx.2008.103986. Epub 2009 Jan 21. PMID 19158125
- [Background] Petros S, Engelmann L. Validity of an abbreviated indirect calorimetry protocol for measurement of resting energy expenditure in mechanically ventilated and spontaneously breathing critically ill patients. Intensive Care Med. 2001 Jul;27(7):1164-8. doi: 10.1007/s001340100941. PMID 11534564
- [Derived] Elizabeth NSH, Yanni T, May LS, Fen TH, Janice LX, Peijun K, Pheng OS, Jie TS, Will LNH. Indirect calorimetry directed feeding and cycling in the older ICU population: a pilot randomised controlled trial. BMC Anesthesiol. 2024 May 7;24(1):171. doi: 10.1186/s12871-024-02507-8. PMID 38714926

DOCUMENTS (1):
  • Study Protocol (2018-02-27): https://cdn.clinicaltrials.gov/large-docs/32/NCT03540732/Prot_000.pdf